CLINICAL TRIAL: NCT03497754
Title: The Use of an External Ultrasound Fixator (ProbeFixR) on Intensive Care Patients, a Feasibility Study. (the Soundprobe Study)
Brief Title: The Use of an External Ultrasound Fixator (ProbeFixR) on Intensive Care Patients
Acronym: Soundprobe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL62664.091.17
Record Dates: First submitted 2017-09-18; First posted 2018-04-13 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Hypovolemia
Keywords: ultrasound; cardiac output; Probefix; passive leg raising test
MeSH Terms: conditions — Hypovolemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Cardiac output measurements (Experimental): Cardiac output will be measured using TTE with and without the use of Probefix so not 2 arms but 2 consecutive measurements in the same patient
  Interventions: Device: Probefix

INTERVENTIONS:
Device: Probefix — A passive leg raising test will be done twice to assess the fluid response. Changes in cardiac output are measured using TTE with and without the use of the Probefix.

SUMMARY:
Study to assess the feasibility of an external ultrasound fixator (ProbeFix)

DETAILED DESCRIPTION:
Rationale: Study to assess the feasibility of an external ultrasound fixator (ProbeFix) Objective: Cardiac output measurements using transthoracic ultrasound (TTE) with and without the use of the probeFixR will be evaluated in terms of accuracy. The TTE measurements will be combined with another form of cardiac output measurements (FlotracR) after a passive leg rasing (PLR) test.

Study design prospective, feasibility study Study population: Adult Intensive Care patients ( > 18 years)

Intervention (if applicable):

Consecutive adult patients on the ICU in which the FlotracR monitor is used will be evaluated after detection of hypovolemia.

Main study parameters/endpoints:

* Percentage of patients in which the ProbeFixR can be used
* The correlation between the measurements done by FlotracR and TTE with and TTE without ProbeFixR

Although no side effects are to be expected the investigators will monitor the patients after the ProbeFix is removed for any skin damage. The investigators will grade this damage into 3 categories:

* No skin marks
* Mild skin marks (no treatment necessary)
* Severe skin marks (surgical or medical treatment necessary)
* If the patients are awake the investigators will ask them whether they felt the ProbeFixR to be unpleasant on a scale of 0-10 (0 being: I did not feel anything and 10 being very unpleasant).

ELIGIBILITY:
Inclusion Criteria:

* Adult Intensive Care patients ( > 18 years), with hypovolemia detected with Flotrac (SVV > 10%)

Exclusion Criteria:

* Pregnancy
* Atrial fibrillation or other irregular heart rhythm
* Pulmonary edema
* PLR not possible (eg neurological disease, spinal trauma, restricted limb movement, deep venous thrombosis, or any other reason as indicated by the attending intensivist).
* age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2019-04-23 (Actual); Study Completion 2019-04-23 (Actual)

PRIMARY OUTCOMES:
The correlation between the measurements done by FlotracR and TTE with and TTE without ProbeFixR | 8 weeks
  A Bland and Altman plot will be constructed and the limits of agreement will be calculated.

SECONDARY OUTCOMES:
Skin marks as possible side effect; scored as 'no skin marks', 'mild skin marks (no treatment necessary)' or 'severe skin marks (surgical or medical treatment necessary)' | 8 weeks
  Percentages will be reported.
Is the Probefix unpleasant on a scale of 0-10 | 8 weeks
  The VAS scale will be reported as mean with standard deviation if normally distributed or as median and inter-quartile range if not normally distributed.
Patients in which the ProbeFixR can be used | 8 weeks
  Percentages will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Bianca Baten, PhD, Study Director — Rijnstate Hospital
Locations (1):
- Rijnstate Hospital, Arnhem, Netherlands

IPD SHARING:
Plan to Share IPD: No